CLINICAL TRIAL: NCT07386938
Title: International, Multicenter, Double-blind, Randomized, Comparative Study of Efficacy, Safety and Pharmacokinetics of RPH-051 and Perjeta® Drug Products Combined With Trastuzumab and Docetaxel as the 1st Line Therapy in Patients With HER2-positive Metastatic or Locally Recurrent Unresectable Breast Cancer
Brief Title: A Study of the Efficacy, Safety and Pharmacokinetics of RPH-051 and Perjeta® in Combination With Trastuzumab and Docetaxel as the 1st Line Therapy in Patients With HER2-positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL011101223
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Locally advanced breast cancer; Metastatic breast cancer; RPH-051
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-051 + Trastuzumab + Docetaxel (Experimental): RPH-051 will be administered on Day 1 of each 21-day cycle, with a loading dose of 840 mg given as a 60-minute intravenous infusion in Cycle 1, followed by a maintenance dose of 420 mg every 3 weeks as a 30-60-minute infusion until disease progression or unacceptable toxicity
  Trastuzumab will be administered on Day 1 of each 21-day cycle, with a loading dose of 8 mg/kg given as a 90-minute intravenous infusion in Cycle 1, followed by a maintenance dose of 6 mg/kg every 3 weeks. If the initial loading dose is well tolerated, trastuzumab may be administered as a 30-minute infusion. Treatment continues until disease progression or unacceptable toxicity
  Docetaxel will be administered on Day 1 of each 21-day cycle at a dose of 75 mg/m^2 for 6 cycles, given as a one-hour intravenous infusion
  Interventions: Drug: RPH-051; Drug: Docetaxel; Drug: Trastuzumab
- Perjeta® + Trastuzumab + Docetaxel (Active Comparator): Perjeta® will be administered on Day 1 of each 21-day cycle, with a loading dose of 840 mg given as a 60-minute intravenous infusion in Cycle 1, followed by a maintenance dose of 420 mg every 3 weeks as a 30-60-minute infusion until disease progression or unacceptable toxicity
  Trastuzumab will be administered on Day 1 of each 21-day cycle, with a loading dose of 8 mg/kg given as a 90-minute intravenous infusion in Cycle 1, followed by a maintenance dose of 6 mg/kg every 3 weeks. If the initial loading dose is well tolerated, trastuzumab may be administered as a 30-minute infusion. Treatment continues until disease progression or unacceptable toxicity
  Docetaxel will be administered on Day 1 of each 21-day cycle at a dose of 75 mg/m^2 for 6 cycles, given as a one-hour intravenous infusion
  Interventions: Drug: Docetaxel; Drug: Perjeta®; Drug: Trastuzumab

INTERVENTIONS:
Drug: RPH-051 — RPH-051: concentrate for solution for infusion, 30 mg/mL
  14 mL of the liquid concentrate is diluted with 250 mL of 0.9% sodium chloride solution. The nominal concentration of the prepared solution is 3.0 mg/mL for the loading dose and 1.6 mg/mL for the maintenance dose
  Arms: RPH-051 + Trastuzumab + Docetaxel
Drug: Docetaxel — Docetaxel: concentrate for solution for infusion, 20 mg/mL
Drug: Perjeta® — Perjeta®: concentrate for solution for infusion, 30 mg/mL
  14 mL of the liquid concentrate is diluted with 250 mL of 0.9% sodium chloride solution. The nominal concentration of the prepared solution is 3.0 mg/mL for the loading dose and 1.6 mg/mL for the maintenance dose
  Arms: Perjeta® + Trastuzumab + Docetaxel
Drug: Trastuzumab — Trastuzumab: lyophilisate for preparation of a concentrate for solution for infusion, 440 mg or 150 mg
  The contents of the vial (440 mg) are dissolved in 20 mL of bacteriostatic water for injection supplied with the drug, containing 1.1% benzyl alcohol. The contents of the vial (150 mg) are dissolved in 7.2 mL of sterile water for injection

SUMMARY:
The main purpose of this study is to prove non-inferiority, as well as to demonstrate the comparability of safety and immunogenicity of RPH-051 and Perjeta® in combination with trastuzumab and docetaxel as the 1st line therapy for patients with HER2-positive breast cancer (BC). Secondary Purposes are to evaluate the pharmacokinetics of RPH-051 in comparison with Perjeta® after a single-dose and repeated intravenous administration

DETAILED DESCRIPTION:
This study is an international, multicenter, double-blind, randomized, comparative, phase III study

Pertuzumab therapy combined with trastuzumab and docetaxel (6 cycles) within this study will last up to 2 years or until the disease progression/development of unacceptable toxicity (whichever comes first)

A subgroup of participants (at least 60 participants, approximately 30 participants in each treatment group) is planned to be included for pharmacokinetic evaluation

The study will include the following periods:

1. Screening period: days -27 to 0 (up to 1 administration of the study therapy)

   If a biopsy of the tumor material to study the HER2 status is required, the screening period can be extended to 42 days
2. Main period: days 1 to 126

   Eligible patients will be randomized at the ratio of 1:1 to one of the two study arms: RPH-051 + trastuzumab + docetaxel or Perjeta® + trastuzumab + docetaxel. On Day 1 (and Day 43 in the PK-subgroup) or the day before, the patients may be hospitalized and will remain in the clinic for up to 24 hours after administration of the first dose of the study drug

   Within the Main period of the Study, the patients will receive pertuzumab (RPH-051 or Perjeta® drug products) combined with trastuzumab and docetaxel according to the following scheme: pertuzumab 420 mg (loading dose 840 mg in the 1st cycle) IV on Day 1 once every 3 weeks + trastuzumab 6 mg/kg (loading dose 8 mg/kg in the 1st cycle) IV on Day 1 once every 3 weeks + docetaxel 75 mg/m2 IV on Day 1 once every 3 weeks, 6 cycles

   In case of significant adverse events (AEs), treatment could be delayed for at least 3 weeks

   The therapy within the Main period will continue until (whichever comes first):
   * 18 weeks (6 cycles)
   * disease progression (according to RECIST 1.1 / clinical progression criteria)
   * development of unacceptable toxicity.
3. Period of extended therapy: days 127 to 365

   During the period of extended therapy, all patients will receive RPH-051 therapy in combination with trastuzumab, including those who received Perjeta® during the Main period. Therapy will be carried out according to the scheme: pertuzumab 420 mg IV once every 3 weeks + trastuzumab 6 mg/kg IV once every 3 weeks

   In case of significant adverse events (AEs), treatment could be delayed for at least 3 weeks

   The therapy during the Period of extended therapy will continue until (whichever comes first):
   * up to 1 year
   * until disease progression (according to RECIST 1.1/clinical progression criteria)
   * development of unacceptable toxicity

   If, after a year of therapy, the patient who achieved control of the disease, she goes into the follow-up care period
4. Follow-up care period: days 366 to 730

   During the follow-up care period, all patients will continue RPH-051 therapy in combination with trastuzumab, including those who received Perjeta® during the Main study period. The therapy will be carried out according to the previous scheme: pertuzumab 420 mg IV once every 3 weeks + trastuzumab 6 mg/kg IV once every 3 weeks

   In case of significant adverse events (AEs), treatment could be delayed for at least 3 weeks

   The therapy during the follow-up care period will continue until (whichever comes first):
   * up to 2 years
   * until disease progression (according to RECIST 1.1/clinical progression criteria)
   * development of unacceptable toxicity
   * the patient's refusal to continue therapy
5. Follow-up period (follow-up/FU)

One follow-up visit (FU-visit) will be scheduled 28 ± 3 days after the last administration

For the patients who early withdraw due to progression of the disease, FU visits will take place once every 6 weeks (counting from the date of the early termination visit) until Day 365 of the study or until lethal outcome

If a patient discontinues the therapy within the main period and the extended therapy period for a reason other than progression of the disease, and other treatment regimen is not prescribed to her, further FU visits will be held in the form of evaluation of the tumor response by CT/MRI once every 6 weeks until Day 126 and then once every 12 weeks until Day 365 of the study or until the disease progression/prescription of other therapy, whichever comes first. Upon the disease progression/prescription of another therapy, the patient follow-up will continue in the form of telephone contacts once every 6 weeks until Study Day 365 or until lethal outcome

If a patient discontinues the therapy with the study drug within the follow-up care period for any reason, FU visits will take place once every 6 weeks (counting from the date of the early termination visit) in the form of telephone contacts until Day 730 of the study or until lethal outcome

ELIGIBILITY:
The patients must meet all the following inclusion criteria:

1. Voluntarily signed and dated Informed Consent Form (ICF) of the patient agreed to take part in this Study
2. Histologically verified (documented results of respective examinations available) metastatic or locally recurrent unresectable breast adenocarcinoma (in case the results of previous examinations are not available, the diagnosis will be verified in the central laboratory during screening upon receipt and evaluation of the results before randomization)
3. Patients with metastatic or locally recurrent unresectable breast cancer (BC) who have indications for the 1st line therapy
4. HER2-positive tumor status, defined as 3+ points according to the results of immunohistochemical examination (IHC) and/or detected amplification of HER2 according to the results of fluorescence in situ hybridization (as defined by a ratio ≥ 2,0), evaluated using a validated test. The HER2 status analysis is carried out in the invasive component of a biopsy sample of tumor tissue during screening in the central laboratory. The results must be obtained before making a decision on randomization of the patient. For analysis, it is required to provide the blocks no more than 1 year old, obtained from the treatment-naive lesions, or a biopsy is performed as a part of screening
5. ECOG status 0-1.
6. Left ventricular ejection fraction (LVEF) ≥ 55 % during the screening.
7. Presence of at least one measurable lesion in accordance with the RECIST 1.1 criteria (if the patient's only measurable lesion is a bone one, she cannot be enrolled in the study).
8. Absence or resolution of the previous therapy toxic effects or negative consequences of surgeries of up to ≤ 1 gr. according to CTCAE 5.0, with the exception of chronic/irreversible adverse events that do not affect the safety parameters of the study therapy (for example, alopecia)
9. Life expectancy of at least 18 weeks from the date of randomization (in the opinion of the Investigator)
10. Consent of a patient with preserved childbearing potential to abstain from heterosexual contact or use reliable methods of contraception, starting from the time the Informed Consent Form is signed, throughout the entire period of treatment within the study and 7 months after receiving the last infusion of pertuzumab and trastuzumab. Female patients are considered to be incapable of childbearing if the final cessation of menstruation is confirmed retrospectively after 12 months of natural amenorrhea, i.e. amenorrhea with an appropriate clinical status, for example, a suitable age

Additional criteria for inclusion in PK subgroups

1. Availability of the signed Informed Consent Form to participate in the pharmacokinetic study
2. Body weight in the range of 40-100 kg at the time the ICF is signed
3. Patient's capability, in the justified opinion of the Investigator, to participate in the pharmacokinetic study and possibility to take the required number of blood samples

The patients cannot be included in the study if any of the following exclusion criteria is met:

1. Previous antitumor therapy for metastatic or locally recurrent unresectable BC (neoadjuvant/adjuvant therapy with trastuzumab and one hormone therapy regimen for the metastatic process are allowed)
2. Previous pertuzumab therapy
3. The period without the signs of disease from the completion of the systemic neoadjuvant or adjuvant BC therapy (except hormonal therapy) to the established diagnosis of the metastatic process or recurrence in < 12 months
4. The period from completion of the systemic neoadjuvant or adjuvant BC therapy with trastuzumab and docetaxel to the start of the systemic therapy for metastatic or locally recurrent unresectable process with a combination of pertuzumab + trastuzumab + docetaxel is < 12 months
5. Sustained hematological toxicity (hemoglobin, leukocytes, neutrophils, platelets) ≥ grade 2, resulting from the previous adjuvant therapy
6. Peripheral neuropathy ≥ grade 3 at the time the ICF is signed
7. Other oncological pathology that is progressing or requires antitumor therapy (including hormonal therapy) within 5 years before signing the ICF, except radically removed cervical carcinoma in situ or radically removed basal cell/squamous cell skin carcinoma
8. Central nervous system metastases that are progressive or accompanied by clinical symptoms (for example, cerebral edema, compression of the spinal cord), or require the application of glucocorticosteroids (GCS) at a dose equivalent to daily intake of prednisolone > 10 mg (or dexamethasone > 1.5 mg), and/or anticonvulsants. Patients with brain metastases can be included in the study if they receive adequate therapy (surgery or radiotherapy) and are stabilized according to the imaging studies data for at least 4 weeks before the expected date of randomization into the study. Patients with CNS metastases detected for the first time as a part of screening, which are not accompanied by neurological symptoms and do not require any therapy, can be included in the study
9. History of treatment with cumulative doses of anthracyclines
10. Patients with severe concomitant diseases, with life-threatening acute complications of the underlying disease
11. Concomitant diseases that are ongoing at the time of the screening examination and that increase the patient's risk of developing adverse events during the application of study therapy:

    * stable effort angina, Functional Class III-IV, unstable angina
    * history of myocardial infarction or stroke occurred less than 6 months before signing of the IC form
    * clinically significant rhythm disturbances (patients with asymptomatic atrial fibrillation can be included in the study provided the ventricular rhythm is controlled)
    * chronic cardiac failure, Class III-IV according to New York Heart Association (NYHA) classification
    * uncontrolled arterial hypertension (systolic blood pressure over 150 mmHg or diastolic blood pressure over 90 mmHg during antihypertensive therapy)
    * decrease in LVEF to < 50 % in the medical history during or after the previous neoadjuvant or adjuvant trastuzumab therapy
    * severe respiratory failure, as well as dyspnea at rest due to complications of advanced cancer or other diseases requiring continuous oxygen therapy
    * current severe uncontrolled systemic disease
    * any other concomitant disease or condition that significantly increases the risk of developing an AE during the study, in the opinion of the Investigator
12. Major surgery or significant injury less than 28 days before, radiation therapy (other than palliative) less than 14 days before the IC form is signed, or a planned major surgery during treatment within this study
13. Non-healing wounds, ulcers at the time the ICF is signed
14. Hematological disorders (in case any of the following):

    * neutrophils < 1.5 x 109/L
    * platelets <100 x 109/L
    * hemoglobin < 90 g/L
15. Renal dysfunction:

    • creatinine > 1.5 × ULN or glomerular filtration rate < 45 mL/min (calculated using CKD-EPI formula)
16. Liver dysfunction (in case any of the following):

    * bilirubin ≥ 1.5 × ULN (except for patients with Gilbert's syndrome, whose total bilirubin values should not exceed 50 µmol/L)
    * AST or ALT ≥ 3 × ULN (5 × ULN for patients with liver metastases)
17. Administration of injectable anticoagulants during the screening period and 3 months before is prohibited. The maximum permissible daily dose of tableted anticoagulants: rivaroxaban - no more than 20 mg, apixaban - no more than 10 mg per day for patients with non-valvular atrial fibrillation and no more than 5 mg for the prevention of recurrence of deep vein thrombosis and/or PATE
18. Conditions that limit the patient's ability to comply with the requirements of the protocol (dementia, neurological or psychiatric disorders, drug addiction, alcohol addiction, religious or personal beliefs of the patient, which may potentially limit standard therapy methods within the study, etc.)
19. Concurrent participation in other interventional and non-interventional clinical studies less than 28 days before the IC form is signed (provided the patient has received at least one dose of experimental therapy), and previous participation in this clinical study (provided the patient has received at least one administration of RPH-051)
20. Current continuous daily treatment with corticosteroids (at a dose equivalent to > 10 mg/day of methylprednisolone) (excluding inhaled steroids)
21. Acute infectious diseases or activation of chronic infectious diseases, including those requiring intravenous injection of antibacterial drugs, less than 28 days before signing of the IC form
22. Active hepatitis B or C, HIV infection, syphilis
23. Inability to administer the study drug intravenously
24. Inability to perform intravenous contrast
25. Hypersensitivity to any of the components of the study drugs specified in the protocol, or intolerance to any of the drug products for premedication
26. Pregnancy or breastfeeding
27. Any other significant concomitant diseases or conditions that could, in the reasonable opinion of the Investigator, adversely affect the patient's participation and well-being in the study and/or distort the evaluation of the study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 246 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (%) (ORR) | Up to day 126
  Objective response rate (%) (ORR) for a period of up to 18 weeks of therapy inclusive. ORR is the percentage of patients in a group achieving either a complete or partial tumor response to therapy. Complete Response (CR) is the disappearance of all target lesions confirmed by the computer tomography (CT) for at least 4 weeks; the short axis of any previously pathological lymph node (target or non-target) must be < 10 mm. Partial Response (PR) is at least a 30% reduction in the sum of diameters of target lesions, maintained for at least 4 weeks compared with baseline (screening) values

SECONDARY OUTCOMES:
Disease control rate (DCR) (%) | Up to day 126
  Disease control rate (DCR) (%) for a period of up to 18 weeks of therapy inclusive. DCR is the percentage of patients in a group achieving a complete or partial tumor response to therapy, or disease stabilization. Stable Disease (SD) is defined as neither a sufficient decrease in the sum of diameters of target lesions to qualify as a partial response, nor an increase in the sum of diameters that would be considered disease progression, compared with the smallest sum of diameters recorded during the observation period
Time to tumor response to therapy (TTR) | Up to day 126
  Time to tumor response to therapy (TTR) for a period of up to 18 weeks of therapy inclusive. TTR is the time from the start of the study therapy to the first documented objective tumor response
Duration of tumor response to therapy (DOR) | Up to day 126
  Duration of tumor response to therapy (DOR) for a period of up to 18 weeks of therapy inclusive. DOR is the time from the first documented objective tumor response to disease progression or death from any cause. Progression (PD) is defined as a ≥20% increase in the sum of diameters of target lesions compared with the smallest sum recorded during the observation period (with an absolute increase of at least 5 mm), or the appearance of one or more new lesions
Progression-free survival (PFS) expressed as PFS level (%) | Up to day 126
  Progression-free survival (PFS) expressed as PFS level (%) for a period of up to 18 weeks of therapy inclusive
Progression-free survival (PFS) expressed as median PFS | Up to day 126
  Progression-free survival (PFS) expressed as median PFS for a period of up to 18 weeks of therapy inclusive
Area under the pharmacokinetic curve "concentration-time" (AUC(0-504)) of pertuzumab | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Area under the pharmacokinetic curve "concentration-time" of pertuzumab after the first (single dose) administration, truncated at the point before the second administration, i.e. up to 504 hours
Maximum serum concentration of pertuzumab after the first administration (Cmax) | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Maximum serum concentration of pertuzumab after the first administration (Cmax)
Maximum serum concentration of pertuzumab at steady state (Cmax ss) after the 3rd administration | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Maximum serum concentration of pertuzumab at steady state (Cmax ss) after the 3rd administration
Minimum serum concentration of pertuzumab at steady state (Cmin ss) after the 3rd administration | Pre-dose immediately before the second, third (Day 43 +2), fourth, fifth (Day 85 +2), and sixth (Day 106 +2) infusions (≤ 30 minutes before administration)
  Minimum serum concentration of pertuzumab at steady state (Cmin ss) after the 3rd administration
Area under the pharmacokinetic curve "concentration-time" of pertuzumab at steady state (AUC tau ss) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Area under the pharmacokinetic curve "concentration-time" of pertuzumab at steady state (AUC tau ss) after the 3rd administration

OTHER OUTCOMES:
Objective response rate (%) (ORR) | Up to day 168
  Objective response rate (%) (ORR) for a period of up to 24 weeks of therapy inclusive
Objective response rate (%) (ORR) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Objective response rate (%) (ORR) for a period of up to 1 year of therapy inclusive (non-comparative evaluation in the RPH-051 group)
Disease control (DCR) (%) | Up to day 168
  Disease control (DCR) (%) for a period of up to 24 weeks of therapy inclusive
Disease control (DCR) (%) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Disease control (DCR) (%) within a period of up to 1 year of therapy inclusive (non-comparative evaluation in the RPH-051 group)
Tumor time to response to therapy (TTR) | Up to day 168
  Tumor time to response to therapy (TTR) for a period of up to 24 weeks of therapy inclusive
Tumor time to response to therapy (TTR) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Tumor time to response to therapy (TTR) within a period of up to 1 year of therapy inclusive (non-comparative evaluation in the RPH-051 group)
Tumor duration to response to therapy (DOR) | Up to day 168
  Tumor duration to response to therapy (DOR) for a period of up to 24 weeks of therapy inclusive
Tumor duration to response to therapy (DOR) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Tumor duration to response to therapy (DOR) within a period of up to 1 year of therapy inclusive (non-comparative evaluation in the RPH-051 group)
Progression-free survival (PFS) (non-comparative evaluation in the RPH-051 group) | Up to day 168
  Progression-free survival (PFS) expressed as the rate (%) of PFS for a period of up to 24 weeks of therapy inclusive
Progression-free survival (PFS) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Progression-free survival (PFS) expressed as the rate (%) of 1-year PFS (non-comparative evaluation in the RPH-051 group)
Progression-free survival (PFS) expressed as median PFS | Up to day 168
  Progression-free survival (PFS) expressed as median PFS for a period of up to 24 weeks of therapy inclusive
Progression-free survival (PFS) expressed as median PFS (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Progression-free survival (PFS) expressed as median PFS for a period of up to 1 year of therapy inclusive (non-comparative evaluation in the RPH-051 group)
Overall survival (OS) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Overall survival (OS) expressed as 1-year OS rate (non-comparative evaluation in the RPH-051 group)
Overall survival (OS) (non-comparative evaluation in the RPH-051 group) | Up to day 365
  Overall survival (OS) expressed as median OS for a period of up to 1 year of therapy (non-comparative evaluation in the RPH-051 group)
Proportion of patients (%) with adverse drug reactions (ADRs) of any severity | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with ADRs of any severity
Proportion of patients (%) with AEs of any severity | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with AEs of any severity
Proportion of patients (%) with AEs of severity grade ≥ 3 | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with AEs of severity grade ≥ 3
Proportion of patients (%) with ADRs of severity grade ≥ 3 | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with ADRs of severity grade ≥ 3
Proportion of patients (%) with serious adverse events (SAEs) | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with SAEs
Proportion of patients (%) with serious adverse drug reactions (SADRs) | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) with SADRs
Proportion of patients (%) who required discontinuation of treatment due to development of ADRs | Days: 1 - 730 (up to 28±2 days after last administration)
  Proportion of patients (%) who required discontinuation of treatment due to development of ADRs
Proportion of patients (%) who developed anti-drug antibodies (ADA) to pertuzumab | Pre-dose on Day 1, 43, 106 (main period) and Day 169, 190, 274, 258 (extended therapy period) (≤ 30 minutes before administration)
  Proportion of patients (%) who developed ADA to pertuzumab
Proportion of patients (%) who developed neutralizing antibodies (NAb) to pertuzumab | Pre-dose on Day 1, 43, 106 (main period) and Day 169, 190, 274, 258 (extended therapy period) (≤ 30 minutes before administration)
  Proportion of patients (%) who developed NAb to pertuzumab
Area under the pharmacokinetic curve "concentration-time" (AUC(0-∞)) of pertuzumab | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Area under the pharmacokinetic curve "concentration-time" of pertuzumab after the first administration to infinity (AUC(0-∞))
Time to reach the maximum concentration of pertuzumab in the blood serum after the first administration (Tmax) | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Time to reach the maximum concentration of pertuzumab in the blood serum after the first administration (Tmax)
Elimination half-life of pertuzumab after the first administration (T1/2) | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Elimination half-life of pertuzumab after the first administration (T1/2)
Volume of distribution of pertuzumab after the first administration (Vd) | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Volume of distribution of pertuzumab after the first administration (Vd)
Elimination rate constant of pertuzumab after the first administration (Kel) | Pre-dose on Day 1 (first administration) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (Day 2), 96 (Day 5), 216 (Day 10), 336 (Day 15), 504 (Day 22) hours post-dose
  Elimination rate constant of pertuzumab after the first administration (Kel)
Area under the pharmacokinetic curve "concentration-time" of pertuzumab to infinity at steady state (AUC(0-∞) ss) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Area under the pharmacokinetic curve "concentration-time" of pertuzumab to infinity at steady state (AUC(0-∞) ss)
Time to reach the maximum concentration of pertuzumab at steady state (Tmax ss) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Time to reach the maximum concentration of pertuzumab at steady state (Tmax ss)
Elimination half-life of pertuzumab at steady state (T1/2 ss) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Elimination half-life of pertuzumab at steady state (T1/2 ss)
Volume of distribution of pertuzumab at steady state (Vd, ss) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Volume of distribution of pertuzumab at steady state (Vd, ss)
Residual concentration of pertuzumab at repeated administration (Cthrough) | Pre-dose on Day 43 (+2 days, third infusion) and 1, 1.5, 2, 2.5, 4, 7, 12 hours post-dose; 24 (+72 h, Day 44 +2), 96 (+72 h, Day 47 +2), 216 (+72 h, Day 52 +2), 336 (+72 h, Day 57 +2), 504 (+72 h, Day 64 +2) hours post-dose
  Residual concentration of pertuzumab at repeated administration (Cthrough)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (45):
- Russia (45):
  - Regional Budgetary Healthcare Institution "Kursk Oncology Research and Clinical Center named after G.E. Ostroverhov", Kursk, Kursk Oblast
  - State Budgetary Healthcare Institution "Leningrad Regional Clinical Hospital" (SBHI "LOKH"), Kuz'molovskiy, Leningradskaya Oblast'
  - State Budgetary Healthcare Institution of Arkhangelsk Region "Arkhangelsk Clinical Oncology Dispensary", Arkhangelsk
  - Regional State Budgetary Healthcare Institution "Altai Regional Oncology Dispensary", Barnaul
  - Private Healthcare Institution "RZD-Medicine Clinical Hospital of Chelyabinsk", Chelyabinsk
  - Regional Budgetary Healthcare Institution "Ivanovo Regional Oncology Dispensary" (RBHI "IvOOD"), Ivanovo
  - State Budgetary Healthcare Institution of Kaluga Region "Kaluga Regional Clinical Oncology Dispensary", Kaluga
  - State Autonomous Healthcare Institution "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigal", Kazan'
  - State Budgetary Healthcare Institution "Kuzbass Clinical Oncology Dispensary named after M.S. Rappoport" (SBHI "KCOD"), Kemerovo
  - Kirov Regional State Clinical Budgetary Healthcare Institution "Center of Oncology and Medical Radiology", Kirov
  - Regional State Budgetary Healthcare Institution "Krasnoyarsk Regional Clinical Oncology Dispensary named after A.I. Kryzhanovsky", Krasnoyarsk
  - State Budgetary Healthcare Institution of the City of Moscow "Moscow Multidisciplinary Clinical Center 'Kommunarka' of the Moscow Department of Healthcare" (SBHI "MMCC 'Kommunarka'"), Moscow
  - Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Autonomous Educational Institution of Higher Education First Moscow State Medical University named after I.M. Sechenov of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Branch of the Limited Liability Company "Hadassah Medical Ltd." (LLC Branch "Hadassah Medical"), Moscow
  - Federal State Autonomous Institution "National Medical Research Center 'Medical and Rehabilitation Center'" of the Ministry of Health of the Russian Federation, Moscow
  - Limited Liability Company "RESEARCH LAB", Moscow
  - State Budgetary Healthcare Institution of the City of Moscow "City Clinical Hospital named after S.S. Yudin" of the Moscow Department of Healthcare, Moscow
  - Joint-Stock Company "Medsi Group of Companies" (JSC "Medsi Group of Companies"), Moscow
  - Federal State Budgetary Institution "N.N. Petrov National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Moscow
  - Private Medical Institution "Euromedservice" (PMI "Euromedservice"), Moscow
  - State Budgetary Healthcare Institution of the City of Moscow "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of the Moscow Department of Healthcare", Moscow
  - Limited Liability Company "Novaya Liniya", Nal'chik
  - State Autonomous Healthcare Institution of the Nizhny Novgorod Region "Research Institute of Clinical Oncology 'Nizhny Novgorod Regional Clinical Oncology Dispensary'", Nizhny Novgorod
  - Limited Liability Company Medical and Sanitary Unit "Clinician-Pretor Clinic", Novosibirsk
  - Federal State Budgetary Institution "National Medical Research Center of Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - Federal State Budgetary Healthcare Institution "Clinical Hospital No. 8 of the Federal Medical-Biological Agency" (FSBHI CH No. 8 FMBA), Obninsk
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk
  - State Budgetary Healthcare Institution of Perm Krai "Perm Krai Oncology Dispensary", Perm
  - State Budgetary Healthcare Institution of Stavropol Krai "Pyatigorsk Interdistrict Oncology Dispensary", Pyatigorsk
  - Federal State Budgetary Institution "National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - Joint-Stock Company "Modern Medical Technologies", Saint Petersburg
  - Limited Liability Company "EuroCityClinic", Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov National Medical Research Center of Oncology" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - State Budgetary Healthcare Institution "St. Petersburg Clinical Scientific and Practical Center for Specialized Medical Care (Oncology) named after N.P. Napalkov", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City Clinical Oncology Dispensary" (SPB SBHI CCOD), Saint Petersburg
  - State Healthcare Institution "Regional Clinical Oncology Dispensary" (SHI "RCOD"), Saratov
  - Regional State Budgetary Healthcare Institution "Smolensk Regional Oncology Clinical Dispensary", Smolensk
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University" of the Ministry of Health of the Russian Federation, Tomsk
  - Federal State Budgetary Scientific Institution "Tomsk National Research Medical Center of the Russian Academy of Sciences" (FSBSI "Tomsk NRMC of the Russian Academy of Sciences"), Tomsk
  - State Healthcare Institution "Tula Regional Clinical Oncology Dispensary" (SHI "TRCOD"), Tula
  - State Autonomous Healthcare Institution "Republican Clinical Oncology Dispensary" of the Ministry of Health of the Republic of Bashkortostan, Ufa
  - State Budgetary Healthcare Institution "Volgograd Regional Clinical Oncology Dispensary", Volgograd
  - State Budgetary Healthcare Institution of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
  - State Autonomous Healthcare Institution of Sverdlovsk Region "Sverdlovsk Regional Oncology Dispensary", Yekaterinburg